CLINICAL TRIAL: NCT03793777
Title: The Effect of Short-term Aronia Melanocarpa Extract Supplementation on Cognitive Function in Healthy Young Adults
Brief Title: The Effect of Aronia Melanocarpa Extract on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: BioActor B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Brainport_002
Record Dates: First submitted 2018-12-19; First posted 2019-01-04 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Function
Keywords: supplementation; cognition; cognitive function; vascular function; microvasculature

STUDY DESIGN:
Intervention Model Description: Cross-over study with 2 intervention conditions
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: block randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): microcrystalline cellulose supplementation
  Interventions: Dietary Supplement: Placebo
- Aronia (Experimental): aronia melanocarpa supplementation
  Interventions: Dietary Supplement: Aronia

INTERVENTIONS:
Dietary Supplement: Aronia — daily supplementation
  Arms: Aronia
Dietary Supplement: Placebo — daily supplementation
  Arms: placebo

SUMMARY:
There is a great interest in improving cognitive performance, including memory and attention. Improved attention is desirable for a large group of people because it is linked to improved performance . Students and professionals can benefit from improved attention and thus performance in academic and other work environments. In addition, cognitive functioning also plays an important role in sports. Various cognitive skills, including attention, reaction time and motor function, have shown that they can influence sport performance. A completely natural supplement with aronia melanocarpa extract could be a promising way to naturally improve cognitive performance.

DETAILED DESCRIPTION:
There is a great interest in improving cognitive performance, including memory and attention. Improved attention is desirable for a large group of people because it is linked to improved performance. Students and professionals can benefit from improved attention and thus performance in academic and other work environments. In addition, cognitive functioning also plays an important role in sports. Various cognitive skills, including attention, reaction time and motor function, have shown that they can influence sport performance. A completely natural supplement with aronia melanocarpa extract could be a promising way to naturally improve cognitive performance. The product in this study is aronia melanocarpa which contains polyphenols. A limited number of clinical studies have already been carried out to see the effect of similar products on cognitive functioning. However, these studies have often been done in older study populations or over a longer period of time. In this study, in healthy adolescents (ages between the 18-35 and with a BMI between 18.5 and 30), the investigators want to test the short term (7 days) effect of aronia melanocarpa extract on cognitive functioning. The investigators will also test the effect of supplementation on the particpant's mood, vascular function, blood biomarkers, retinal vasculature, and subjective cognition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults: ages between 18 and 35
* BM between 18.5-30 kg/m2

Exclusion Criteria:

* Current use of (antioxidant) dietary supplements and not willing to quit for the duration of the study duration
* Pre-existing or history of neurological illness
* High blood pressure (>140 systolic and/or >90 diastolic mmHg)
* Use of medication that might have influence on endpoints (e.g. antidepressant)
* Known pregnancy or lactation
* Food allergy to the study product
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study, to be decided by the principle investigator, in the 180 days prior to the study
* Abuse of products (> 20 alcoholic consumptions per week and drug usage)
* Participation in a scientific intervention study which may interfere with this study in the 180 days prior to this study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Cognitive function | After 7 days of supplementation
  CANTAB

SECONDARY OUTCOMES:
Mood | After 7 days of supplementation
  VAMS
Biomarkers in blood and saliva | After 7 days of supplementation
  BDNF & cortisol
Vascular function | After 7 days of supplementation
  SBP & DBP, PWA & PWV
Microvasculature | After 7 days of supplementation
  Fundus photography
Subjective cognition | After 7 days of supplementation
  Cognitive Failures Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahles S, Joris PJ, Plat J. Short-term Aronia melanocarpa extract supplementation improves cognitive performance: a randomized, double-blind, placebo-controlled cross-over study in healthy young adults. Eur J Nutr. 2024 Aug;63(5):1545-1553. doi: 10.1007/s00394-024-03381-3. Epub 2024 Apr 24. PMID 38656355